CLINICAL TRIAL: NCT00865579
Title: Open-Label Trial to Determine the Long-Term Safety of Safinamide in Parkinson's Disease Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: study terminated early due to change in Sponsorship
Sponsor: Newron Pharmaceuticals SPA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 28850; 63,901; EudraCT-Number: 2008-005492-94
Record Dates: First submitted 2009-03-10; First posted 2009-03-19 (Estimated); Last update posted 2017-09-18 (Actual); Status verified 2017-09

CONDITIONS: Parkinson's Disease
Keywords: MAO inhibitors; motor fluctuations; dyskinesia; Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease; Dyskinesias | interventions — safinamide

ARMS (1):
- 1 (Experimental): All subjects to receive first 50mg/d Safinamide with an increase of target dose of 100mg/d after 14 days of taper period until end of treatment visit. In case of any intolerance the daily dose of 100mg might be decreased to 50mg/d. Patients permanently discontinuing treatment will enter a 7day taper phase before treatment discontinuation at a dose of 50mg/day. Subjects already taking 50mg/d may stop Safinamide immediately.
  Interventions: Drug: Safinamide

INTERVENTIONS:
Drug: Safinamide — The Investigational Medicinal Product will be provided by the Sponsor in the form of tablets at dosage strengths of safinamide 50 mg (small - 7 mm) or safinamide 100 mg (large - 9 mm).
  Trial Medication is to be taken once daily, in the morning.

SUMMARY:
Parkinson's Disease (PD) is a major neurodegenerative disorder in which there is a progressive loss of dopamine-containing neurons. The understanding that PD is a syndrome of dopamine (DA) deficiency led to the introduction in the clinical practice of L-dopa, a precursor of DA that crosses the blood brain barrier, and also to the use of selective inhibitors of MAO-B, the major DA metabolising enzyme in humans.

Safinamide is an inhibitor of MAO-B. This study is to evaluate the long term safety and tolerability of safinamide in PD patients, that have already completed a previous clinical study with Safinamide. The physical and neurological conditions as well as other safety parameters will get compared from baseline to subsequent visits.

ELIGIBILITY:
Inclusion Criteria:

1. the subject has completed a previous clinical study with Safinamide in PD
2. the subject successfully completed all trial requirements of the antecedent trial
3. if female, they must be either post-menopausal for at least 2 years, surgically sterilized or have undergone hysterectomy or, if of child bearing potential, they must be willing to avoid pregnancy by using an adequate method of contraception for four weeks prior to, during and four weeks after the last dose of study medication. For the purpose of this trial women of child bearing potential are defined of all female subjects after puberty unless they are postmenopausal for at least two years, are surgically sterile or are sexually inactive
4. subjects must be willing and able to participate in the trial and provide written informed consent

Exclusion Criteria:

1. the subject experienced a clinically significant adverse effect to attributable to Investigational Medicinal Product (IMP) during a previous trial that could put the subject at risk for further treatment with Safinamide
2. if female, the subject is pregnant or lactating
3. any medical issues, which have emerged since the initial clinical trial, that in the opinion of the investigator precludes a subject's ability to participate in this open-label trial

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 964 (Actual)
Dates: Start 2009-04 (Actual); Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Physical Exams | Anticipated time frame up to 3 years
Change from baseline in Neurologic Exams | Anticipated time frame up to 3 years
Change from baseline in Vital Signs | Anticipated time frame up to 3 years
Change from baseline in Laboratory Evaluations | Anticipated time frame up to 3 years
Change from baseline in Electrocardiograms | Anticipated time frame up to 3 years
Summary of Participants who had Adverse Experiences | Anticipated time frame up to 3 years
Change from baseline in Unified Parkinson's Disease Rating Scale (UPDRS) | Anticipated time frame up to 3 years
Change from baseline in Dermatologic Exams | Anticipated time frame up to 3 years
Change from baseline in Ophthalmologic Exams | Anticipated time frame up to 3 years

SECONDARY OUTCOMES:
Change from baseline in Health Resource Utilisation | Anticipated time frame up to 3 years
Change from baseline in EuroQol Group EQ-5D™ Quality of Life Scale | Anticipated time frame up to 3 years
Change from baseline in Parkinson Disease Questionnaire 39 (PDQ-39) | Anticipated time frame up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Willmer, MD, Study Director — EMD Serono Inc., an Affiliate of Merck KGaA, Darmstadt, Germany
Locations (1):
- Research Site, Timuș, Romania

IPD SHARING:
Plan to Share IPD: No
No efficacy endpoints were analyzed in this trial.